CLINICAL TRIAL: NCT06452030
Title: Changing Trunk Muscle Activation in Patients With Recurrent Low Back Pain in Remission
Acronym: MAS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: VZW Educatieve Lichaamsbeweging (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ONZ-2022-0310
Record Dates: First submitted 2024-04-11; First posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Recurrent Low Back Pain; Remission
Keywords: Low back pain; Motor control; Exercise; Randomised Controlled Trial
MeSH Terms: conditions — Low Back Pain; Motor Activity

STUDY DESIGN:
Intervention Model Description: The study model is parallel. Participants with recurrent low back pain in remission will be randomly allocated to receive either (1) specific sensorimotor control training, (2) general extension training or (3) fascia therapy (i.e. parallel study model).
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Specific sensorimotor control training (Experimental): One low-load treatment session of selective multifidus activation.
  Interventions: Behavioral: Specific sensorimotor control training
- Aspecific extension training (Active Comparator): One low-load treatment session of back muscle activation.
  Interventions: Behavioral: Aspecific extension training
- Fascia training (Experimental): One low-load treatment session of general movement exercises.
  Interventions: Behavioral: Fascia training

INTERVENTIONS:
Behavioral: Specific sensorimotor control training — Participants allocated to the specific motor control group will receive sensorimotor training of the multifidus muscle.
  Arms: Specific sensorimotor control training
Behavioral: Aspecific extension training — Participants allocated to the aspecific group will receive spinal extension exercises.
  Arms: Aspecific extension training
Behavioral: Fascia training — Participants allocated to the fascia group will receive general movement exercises.
  Arms: Fascia training

SUMMARY:
The first aim of the study is to investigate the effects of a single therapy session on trunk muscle activation and lumbopelvic sensorimotor control in persons with recurrent low back pain in remission.

The second aim of the study is to examine the convergent validity of (in)voluntary multifidus activation by means of inspection and palpation during two clinically assessed lumbopelvic sensorimotor control tests in persons with recurrent low back pain in remission. The convergent validity will be examined by calculating the relationship between (1) the clinical score of (in)voluntary multifidus activation, (2) back muscle activation during the same tests measured simultaneously with electromyography and (3) trunk muscle activation during other functional movements measured with electromyography.

The third aim of the study is to investigate the convergent validity of a left-right discrimination test by calculating the relationship between (1) the left-right discrimination test, (2) position-reposition test, (3) the Fremantle Back Awareness Questionnaire and (4) the Photograph Series of Daily Activities Scale.

DETAILED DESCRIPTION:
Low back pain (LBP) is a very common musculoskeletal disorder. Previous research has already demonstrated that trunk muscle function and sensorimotor control (SMC) are altered in people with LBP, which may be an important underlying mechanism contributing to their pain. While there is some evidence regarding the immediate effects of exercise therapy on back muscle function (i.e., earlier onset of activity after one therapy session), the effects of a single therapy session on functional movements and clinically assessed SMC tests in patients with recurrent LBP in remission have never been investigated.

Inspection and palpation are often used in clinical settings to detect lumbopelvic SMC changes in people with LBP. If lumbopelvic SMC changes are noted during the clinical examination, specific SMC therapy can be implemented into the treatment plan. Thus, it is critical that the clinically assessed lumbopelvic SMC tests are sufficiently valid. An important prerequisite is that the clinically assessed SMC parameter is related to objectively measured SMC parameters during the same test. However, clinically assessed lumbopelvic SMC tests are often performed in standardized and less functional positions (e.g., prone lying). As such, the question arises whether results from clinically assessed SMC tests are associated with objective SMC parameters evaluated during functional activities relevant for the individual patient (e.g., lifting). Our systematic review showed that only one clinically assessed lumbopelvic SMC test had sufficient convergent validity with low quality of evidence (Brandt et al., 2024). Moreover, no studies investigated the relationships between clinically assessed lumbopelvic SMC tests and objectively measured SMC parameters during a functional task. Further high-quality studies are therefore needed.

In addition, the left-right discrimination test is also accessible in clinical settings. The left-right discrimination test assesses a person's body perception. During this test, the participant must view images on a computer of a person with the trunk flexed or rotated to the left or right. The participant must indicate as quickly and accurately as possible which side of the trunk of the person in the image is bent or turned. Another way to assess body perception is by using the Fremantle Back Awareness Questionnaire, of which the Dutch version was recently validated. It has been suggested that body perception is the result of the interaction of internal "body maps," sensory information, motor output, and beliefs and perceptions about the body. However, the relationship between the left-right discrimination test, the position-reposition test, and the Fremantle Back Awareness Questionnaire has not yet been explored.

ELIGIBILITY:
Inclusion Criteria:

1. People between 18-65 years old
2. Having recurrent non-specific low back pain (LBP) in remission at enrolment:

   * At least 2 episodes of LBP/year, with an 'episode' implying pain lasting a minimum of 24 hours which is preceded and followed by at least 1 month without LBP
   * Minimum LBP intensity during episodes should be ≥2/10 on a numeric rating scale (NRS) from 0 to 10
   * During remission the NRS intensity for LBP should be 0-1/10.
3. Having a dominant flexion movement pattern/ neutral movement pattern

Exclusion Criteria:

1. People <18 years old or >65 years old
2. Having any other type of non-specific LBP (acute, subacute, chronic).
3. Having an active extension movement pattern
4. Having any type of blood clotting disorder
5. People with upper-limb complaints that prevent them from exerting (maximum) force with their arms or hands.
6. People that received specific sensorimotor control training or fascia-training in the previous year
7. People with serious underlying conditions (e.g., multiple sclerosis) or severe scoliosis
8. People with a history of spine surgery
9. Pregnant women and women who have given birth in the year before enrolment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2024-03-29 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Trunk muscle onset during the rapid arm movement test | Baseline
  Trunk muscle onset latencies in response to the unilateral rapid arm movement test will be measured by means of electromyography.
Trunk muscle onset during the rapid arm movement test | Immediately after therapy
  Trunk muscle onset latencies in response to the unilateral rapid arm movement test will be measured by means of electromyography.

SECONDARY OUTCOMES:
Trunk muscle (co-)activation | Baseline
  The participant sits on a stool and holds a horizontal bar with both hands, shoulders at 90 degrees (arms are horizontal). The horizontal bar is secured to the ground using a rope and weights. The participant pushes the horizontal bar upwards without moving the arms, pelvis, or spine. The activation of the back and abdominal muscles will be further investigated.
Trunk muscle (co-)activation | Immediately after therapy
  The participant sits on a stool and holds a horizontal bar with both hands, shoulders at 90 degrees (arms are horizontal). The horizontal bar is secured to the ground using a rope and weights. The participant pushes the horizontal bar upwards without moving the arms, pelvis, or spine. The activation of the back and abdominal muscles will be further investigated.
Back muscle activation | Baseline
  Back muscle activation will be analyzed during (1) bilateral reaching in standing position, (2) bilateral reaching starting in neutral sitting position, and (3) bilateral reaching starting in habitual sitting position.
Back muscle activation | Immediately after therapy
  Back muscle activation will be analyzed during (1) bilateral reaching in standing position, (2) bilateral reaching starting in neutral sitting position, and (3) bilateral reaching starting in habitual sitting position.
Voluntary multifidus activation | Baseline
  Voluntary multifidus activation will be measured while the participant lies prone on a treatment table. The participant will be instructed to gently activate the multifidus muscle without movement of the pelvis or spine, while breathing is maintained.
Voluntary multifidus activation | Immediately after therapy
  Voluntary multifidus activation will be measured while the participant lies prone on a treatment table. The participant will be instructed to gently activate the multifidus muscle without movement of the pelvis or spine, while breathing is maintained.
Involuntary multifidus activation | Baseline
  Involuntary multifidus activation will be assessed by means of the multifidus lift test (Hebert et al., 2015). The participant is lying in the prone position with the shoulders in 120° abduction and 90° flexion at the elbows. The participant will be asked to lift the entire arm approximately 5 cm from the treatment table. The multifidus activation on the contralateral side will be investigated further.
Involuntary multifidus activation | Immediately after therapy
  Involuntary multifidus activation will be assessed by means of the multifidus lift test (Hebert et al., 2015). The participant is lying in the prone position with the shoulders in 120° abduction and 90° flexion at the elbows. The participant will be asked to lift the entire arm approximately 5 cm from the treatment table. The multifidus activation on the contralateral side will be investigated further.
Lumbar proprioception | Baseline
  Lumbar proprioception will be evaluated by means of the position-reposition test. First, the spine of the participant spine is placed in a reference position (50% of maximum range of motion). Second, the participant is asked to return to a neutral sitting position and then to resume the reference position (50% of maximum range of motion). The difference between the two positions will be further investigated.
Left-right discrimination test | Baseline
  During the left-right discrimination test, the participants are required to view images on a tablet of a person whose trunk is bent or rotated to the left or right. The participant must press 'left' or 'right' as quickly and accurately as possible to indicate which side the person's trunk on the image is bent or rotated. The accuracy and speed will be further analyzed.
Disability (questionnaire) | Baseline
  The Roland Morris Disability Questionnaire will be used to evaluate disability.
Body perception (questionnaire) | Baseline
  The Fremantle Back Awareness Questionnaire will be used to evaluate body perception.
Kinesiophobia | Baseline
  The Tampa Scale for Kinesiophobia will be used to evaluate kinesiophobia.
Perceived harmfulness | Baseline
  The Photograph Series of Daily Activities will be used to evaluate perceived harmfulness.

CONTACTS AND LOCATIONS:
Overall Officials: Lieven Danneels, Prof, Principal Investigator — University Ghent
Locations (1):
- Ghent University, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Vet HC, Heymans MW, Dunn KM, Pope DP, van der Beek AJ, Macfarlane GJ, Bouter LM, Croft PR. Episodes of low back pain: a proposal for uniform definitions to be used in research. Spine (Phila Pa 1976). 2002 Nov 1;27(21):2409-16. doi: 10.1097/01.BRS.0000030307.34002.BE. PMID 12438991
- [Background] Stanton TR, Latimer J, Maher CG, Hancock MJ. A modified Delphi approach to standardize low back pain recurrence terminology. Eur Spine J. 2011 May;20(5):744-52. doi: 10.1007/s00586-010-1671-8. Epub 2010 Dec 31. PMID 21193932
- [Background] Tsao H, Hodges PW. Immediate changes in feedforward postural adjustments following voluntary motor training. Exp Brain Res. 2007 Aug;181(4):537-46. doi: 10.1007/s00221-007-0950-z. Epub 2007 May 3. PMID 17476489
- [Background] Tsao H, Druitt TR, Schollum TM, Hodges PW. Motor training of the lumbar paraspinal muscles induces immediate changes in motor coordination in patients with recurrent low back pain. J Pain. 2010 Nov;11(11):1120-8. doi: 10.1016/j.jpain.2010.02.004. PMID 20434958
- [Background] Matheve T, Hodges P, Danneels L. The Role of Back Muscle Dysfunctions in Chronic Low Back Pain: State-of-the-Art and Clinical Implications. J Clin Med. 2023 Aug 24;12(17):5510. doi: 10.3390/jcm12175510. PMID 37685576
- [Background] Hodges PW, Danneels L. Changes in Structure and Function of the Back Muscles in Low Back Pain: Different Time Points, Observations, and Mechanisms. J Orthop Sports Phys Ther. 2019 Jun;49(6):464-476. doi: 10.2519/jospt.2019.8827. PMID 31151377
- [Background] Hebert JJ, Koppenhaver SL, Teyhen DS, Walker BF, Fritz JM. The evaluation of lumbar multifidus muscle function via palpation: reliability and validity of a new clinical test. Spine J. 2015 Jun 1;15(6):1196-202. doi: 10.1016/j.spinee.2013.08.056. Epub 2013 Oct 4. PMID 24314767
- [Background] Meier R, Iten P, Luomajoki H. Clinical assessments can discriminate altered body perception in patients with unilateral chronic low back pain, but not differences between affected and unaffected side. Musculoskelet Sci Pract. 2019 Feb;39:136-143. doi: 10.1016/j.msksp.2018.12.006. Epub 2018 Dec 21. PMID 30593940
- [Background] Brandt M, Danneels L, Meirezonne H, Van Oosterwijck J, Willems T, Matheve T. Clinically assessed lumbopelvic sensorimotor control tests in low back pain: are they actually valid? A systematic review according to COSMIN guidelines. Musculoskelet Sci Pract. 2024 Jun;71:102953. doi: 10.1016/j.msksp.2024.102953. Epub 2024 Apr 7. PMID 38604022